CLINICAL TRIAL: NCT05374889
Title: The Effect of Open Kinetic Chain Proprioception Exercises on Joint Position Sense, Stability, Endurance and Strength in Adolescent Basketball Players
Brief Title: Evaluation of the Contribution of Basketball-specific Target Shooting Exercises to Strength, Position Sense, Stability and Endurance in Young Basketball Players
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Gulsum Mandir Comert, Principal Investigator, Istanbul University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2020/220
Record Dates: First submitted 2022-05-04; First posted 2022-05-16 (Actual); Last update posted 2022-05-16 (Actual); Status verified 2022-05

CONDITIONS: Open Kinetic Chain Proprioception Exercises
Keywords: Proprioception; strength; stability; endurance; adolescent basketball player

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise Group (Experimental): Athletes were asked to throw the ball at predetermined targets in different positions with their eyes closed. In the first exercise, the athlete was positioned 2 m from the target in a sitting position, facing the marked lines on the wall. It was asked to make 3 trial shots with a basketball ball while the eyes were open, from the bottom up to the 3 lines on the wall. Then the shots were made while the eyes were closed. In the next exercise, it was requested to make 3 trial shots from the bottom up by looking at the same 3 lines marked in the supine position at the distance of 1 m from the target. Then the shots were made with the eyes facing the ceiling. The last exercise was in a standing position, from the line marked 5 m from the target to the basket, it was requested to make 3 trial free throw with eyes open to the basket. Then, after each throw, the athlete was asked to turn around his own axis and continue to next throw, with eyes closed.
  Interventions: Other: Open Kinetic Chain Proprioception Exercises
- Control Group (No Intervention): Control group did not participate in any exercise program.

INTERVENTIONS:
Other: Open Kinetic Chain Proprioception Exercises — basketball-specific target shooting in open kinetic chain
  Arms: Exercise Group

SUMMARY:
The aim of this study is to examine the effects of open kinetic chain proprioception exercises on joint position sense, strength, functional stability and endurance in adolescent basketball players

DETAILED DESCRIPTION:
Adolescent basketball players, aged 13-16, were randomly divided into two groups as exercise group (n = 11) and control group (n = 11). Exercise group performed open kinetic chain functional proprioception exercises twice a week for 6 weeks. Control group did not participate in any exercise program. Before and after the exercise program all athletes were subjected to the proprioception test and isokinetic muscle strength test on the isokinetic dynamometer, closed kinetic chain upper extremity stability test and modified push-up test.

ELIGIBILITY:
Inclusion Criteria:

* being 13-16 years old
* being male
* playing basketball regularly

Exclusion Criteria:

* having any upper extremity muscle injury in the last 6 months,
* having a limitation in the shoulder girdle range of motion,
* having a shoulder, elbow, wrist dislocation problems

Ages: 13 Years to 16 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 22 (Actual)
Dates: Start 2020-01-02 (Actual); Primary Completion 2020-03-15 (Actual); Study Completion 2020-06-20 (Actual)

PRIMARY OUTCOMES:
Proprioception test- Cybex-Humac NORM | 20 minutes
  Position-based proprioception test with Cybex-Humac NORM in 60 ̊ and 120 ̊ angles
Peak Torque & Peak Torque/Body Weight- Cybex-Humac NORM | 20 minutes
  Strength and endurance tests with Cybex-Humac NORM at 60°/sec and 180°/sec angular velocities
Closed kinetic chain upper extremity stability test | 5 minutes
  Recording the number of touches in 15 seconds
Modified push-up test | 10 minutes
  Recording the number of push-ups

CONTACTS AND LOCATIONS:
Overall Officials: Gulsum Mandir Comert, M.Sc., Principal Investigator — Istanbul University
Locations (1):
- Istanbul Faculty of Medicine, Sports Medicine Department, Istanbul, Turkey (Türkiye)